CLINICAL TRIAL: NCT06174805
Title: A Prospective Multi-Center, Single-Arm Study of Endoscopic Ultrasound-Guided Gastroenterostomy With Lumen-Apposing Metal Stent for Gastric Outlet Obstruction From Malignant Unresectable Disease
Brief Title: AXIOS™ Gastroenterostomy for Gastric Outlet Obstruction IDE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7152
Record Dates: First submitted 2023-12-04; First posted 2023-12-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Gastric Outlet Obstruction
Keywords: GOO; Gastric Outlet Obstruction; AXIOS; Gastroenterostomy
MeSH Terms: conditions — Gastric Outlet Obstruction | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AXIOS(TM) Stent and Electrocautery Enhanced Delivery System (Experimental): Patients who meet all the inclusion criteria and none of the exclusion criteria will have a EUS-guided gastroenterostomy (EUS-GE) using the AXIOS(TM) lumen-apposing Metal Stent for the management of symptoms associated with gastric outlet obstruction from malignant unresectable neoplasm
  Interventions: Device: AXIOS(TM) Stent and Electrocautery Enhanced Delivery System

INTERVENTIONS:
Device: AXIOS(TM) Stent and Electrocautery Enhanced Delivery System — Patients who meet all the inclusion criteria and none of the exclusion criteria will have a EUS-guided gastroenterostomy (EUS-GE) using the AXIOS(TM) lumen-apposing Metal Stent for the management of symptoms associated with gastric outlet obstruction from malignant unresectable neoplasm

SUMMARY:
To investigate the safety and technical success of EUS-guided gastroenterostomy (EUS-GE) using the AXIOSTM lumen-apposing Metal Stent for the management of symptoms associated with gastric outlet obstruction from malignant unresectable neoplasm.

DETAILED DESCRIPTION:
The study is a prospective multi-center, single -arm study with treatment of up to 67 subjects at up to 10 clinical centers. Subjects who meet all eligibility criteria will receive the AXIOS stent and up to 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Gastric outlet obstruction from unresectable malignant neoplasm
2. Eligible for endoscopic intervention
3. GOOS of 0 or 1 0 - no oral intake 1 - liquids only 2 - soft solids only 3 - low-residue or full diet
4. 18 years of age or older
5. Willing and able to comply with the study procedures or legally authorized representative (LAR) must provide written informed consent form (ICF) to participate in the study
6. The distance between the gastric lumen and jejunal lumen must be no more than 1.0 cm

Exclusion Criteria:

1. Patients with baseline ECOG > 2 and/or Karnofsky Performance score < 30
2. Gastric cancer or any malignant infiltration precluding a cancer free puncture site of the AXIOSTM stent
3. Abnormal coagulation INR > 1.5 and not correctable (per the discretion of the physician) or who require continuous complete anticoagulation, and/or any underlying condition associated with high risk of bleeding
4. Altered anatomy of the upper gastrointestinal tract due to surgery of esophagus, stomach and duodenum that might preclude endoscopic gastroenterostomy
5. Multiple-level bowel obstruction downstream from the intended location of the EUS-guided bypass confirmed by radiography such as small bowel series or computed tomography
6. Presence of intraperitoneal fat between the gastric lumen and jejunal lumen estimated to be larger than 1.0 cm at the proposed site of AXIOSTM stent insertion
7. Gastric varices located within a two-centimeter radius of the device insertion location on the gastric wall
8. Ascites Grade ≥ 2 confirmed by cross-sectional imaging
9. Vessels located within a two-centimeter radius of the device insertion location
10. History of multiple abdominal surgeries and/or evidence of small bowel adhesions
11. Allergic to any of the device materials
12. Contraindications to use of electrical devices
13. Pregnancy
14. Prisoners and other vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Through study completion, an average of 1 year
  AXIOS stent related or AXIOS endoscopic and/or study procedure related serious adverse events through 30 days post stent placement.
Primary Technical Success Endpoint | During the procedure
  Successful stent placement, defined as transmural placement of the AXIOS stent with confirmed stent patency by visualization of the contralateral wall of the small bowel through the AXIOS stent lumen. Visualization of blue dye in the gastric lumen or injection of contrast to confirm continuity of the gastroenteric lumen, may be used to provide supplemental confirmation of intended stent placement. Note: Visualization of blue dye in the gastric lumen or injection of contrast to confirm continuity of the gastroenteric lumen, may be used to provide supplemental confirmation of intended stent placement.
Primary Effectiveness Endpoint | through 14 days after procedure
  Clinical Success defined as improvement of Gastric Outlet Obstruction Score (GOOS)by 1 point from baseline to any point during 14 days after AXIOS stent placement and GOOS remaining at 1 or more without the need for reintervention due to loss of stent function at 30 days post-index procedure or death, whichever comes first.

OTHER OUTCOMES:
Clinical success over time defined as improvement of GOOS by 1 point from baseline at any time during 14 days after AXIOS stent placement and GOOS remaining at 1 or more. This endpoint will be evaluated at 3 months, 6 months, and 12 months | Through study completion, an average of 1 year
  A patient undergoing reintervention for GOO is considered a failure of clinical success
Time to resumption of oral intake after stent placement. | Immediately after the procedure
Time to start or resume chemotherapy after AXIOSTM stent placement (where applicable) | Immediately after the procedure
Change in Quality-of-Life score (SF-12 questionnaire) from baseline to 30 days, 3 months, 6 months, and 12 months | Through study completion, an average of 1 year
Incidence of Device Deficiencies | Immediately after the procedure
  Including but not limited to stent migration/misplacement, stent occlusion, leakage at site of stent placement.
Incidence of Reintervention for GOO | Immediately after the procedure
  defined as need for repeat treatment for persistent or recurrent GOO symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shayan Irani, MBBS, MD, Principal Investigator — Virginia Mason Medical Center
Locations (10):
- United States (5):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian/ Weill Cornell Medical Center, New York, New York
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
- UZ Leuven, Leuven, Belgium
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, Brazil
- McGill University Health Care, Montreal, Canada
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China
- Asian Institute of Gastroenterology, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Undecided